CLINICAL TRIAL: NCT07188168
Title: Objective Assessment of Tooth Mobility Using the Osstell Device: A Custom-Bonded Apparatus Trial
Brief Title: Assessment of Tooth Mobility Using the Osstell Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Osman Fatih Arpag, Head of the Oral and Dental Health Hospital, Mustafa Kemal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022/35 (Ethical number)
Record Dates: First submitted 2025-09-07; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Tooth Mobility
Keywords: resonance frequency analysis; periotest; Miller mobility index
MeSH Terms: conditions — Tooth Mobility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobility group (Other): The participants' mobile teeth were assessed using three different tooth mobility measurement methods, and the agreement among these measurements was evaluated.
  Interventions: Device: Miller mobility measurement

INTERVENTIONS:
Device: Miller mobility measurement — Tooth mobility at different levels of mobility was assessed using Miller, Periotest and Osstell, and was evaluated both subjectively and objectively.
  Other Names: Periotest; Osstell Beacon

SUMMARY:
In this trial, it is hypothesized that mobility values obtained from natural teeth using the Osstell device-adapted with a specifically designed attachment-will demonstrate a statistically significant correlation with those obtained through established methods such as the Periotest and the Miller index. Accordingly, the aim of this study is to investigate the applicability of the Osstell device for assessing the mobility of natural teeth having different mobility grades and to evaluate the correlation between its measurements and those derived from conventional clinical mobility assessment methods.

DETAILED DESCRIPTION:
A total of 16 patients, including 10 males and 6 females, were selected for the study, and mobility measurements were performed on 94 permanent teeth. All measurements were performed twice on each tooth by the same calibrated investigator to ensure consistency and eliminate inter-examiner variability. The repeated measurements were carried out under identical conditions for each assessment method (Miller mobility grading, Periotest M, and Osstell Beacon). To evaluate the intra-examiner reliability, the agreement of the two consecutive measurements was assessed using appropriate statistical methods. High intra-examiner agreement was considered indicative of the measurement reliability and reproducibility within the study. To assess tooth stability, resonance frequency analysis was performed using the Osstell Beacon device (Osstell, AB, Gothenburg, Sweden).

A custom-fabricated titanium bracket was used to accommodate the smartPeg and ensure standardized placement on each tooth. The bracket-like apparatus was carefully aligned with the long axis of the tooth and positioned apically.

Bracket specifications

* Raw material: Medical-grade titanium, precision-machined using Computer Numerical Control technology.
* Design: Cylindrical base with a centrally located, threaded slot for smartPeg insertion SmartPeg thread slot
* Internally threaded to enable clockwise insertion of the smartPeg (Figures 3b and 3c)
* Thread type: micro-thread,
* Tapered, centred aperture
* Diameter: approximately 1.2-1.5 mm Tooth contact surface
* Flat base designed to conform to the buccal surface of the tooth
* Smooth texture with micro-mechanical retention properties
* Suitable for adhesive fixation or direct contact application The apparatus was placed on the buccal surface of the respective tooth using flowable composite. Care was taken to ensure that the slot of the bracket designated for a smartPeg placement was oriented toward the root. Subsequently, the smartPeg was positioned in alignment with the root and torqued into place. After the smartPeg installation, two measurements were taken from different directions. The mean of the two readings was recorded as the final RFA value for each tooth. The Osstell Beacon was operated at a 2-5 mm distance, held perpendicular (90°) to the smartPeg without making contact. In this approach, the unit of measurement is the Implant Stability Quotient (ISQ), which is derived from resonance frequency analysis and ranges from 0 to 100, with higher values indicating greater stiffness at the implant-bone interface.The normality of the data distribution was tested using the Shapiro-Wilk test. The relationships between numerical variables were evaluated using Spearman's correlation coefficient. To assess the agreement between mobility classes and the Periotest and Osstell groups, Cohen's Kappa statistic was employed. The Kappa coefficient was interpreted as follows: values <0.00 indicated "poor agreement," 0.00-0.20 "slight agreement," 0.21-0.40 "fair agreement," 0.41-0.60 "moderate agreement," 0.61-0.80 "substantial agreement," and 0.81-1.00 "almost perfect agreement." The reliability of stability scores obtained from the Periotest and Osstell devices was evaluated using the Intraclass Correlation Coefficient (ICC). To determine inter-device agreement, ICC values were calculated based on a two-way mixed-effects model using the single measurement (average measure) approach. ICC values ≥0.75 were considered to indicate satisfactory reliability. All statistical analyses were performed using SPSS (Statistical Package for the Social Sciences), with a significance level set at 5% (p<0.05)

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 45 years.
* Systemically healthy individuals
* Teeth which they have intact periodontium or treated because of periodontal disease.

Exclusion Criteria:

* History of psychiatric or neurological disorders.
* Impaired muscle coordination or neuromuscular dysfunction.
* Patients undergoing orthodontic treatment or with recent dental trauma affecting tooth stability.
* Presence of parafunctional habits such as bruxism (teeth grinding) or clenching.
* Presence of tooth pathologies such as endodontic or root resorption.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Miller measurement | Baseline (first day)
  Tooth mobility was classified from 0 to 3 according to the Miller index.
Periotest measurements | Baseline (first day)
  Tooth mobility was measured using the Periotest device, with values ranging from -8 to +50.
Osstell Measuements | Baseline (first day)
  Tooth resonance frequency was assessed using the Osstell device, and the values were classified as less than 60, between 60 and 69, and greater than 69.

CONTACTS AND LOCATIONS:
Overall Officials: Fariz Selimli, Assoc Prof, Study Director — Mustafa Kemal University
Locations (1):
- Hatay Mustafa Kemal University, Antakya, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No